CLINICAL TRIAL: NCT04629170
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Assess the Safety, Tolerability, and Pharmacodynamics of SYNB8802 in Healthy Volunteers and in Patients With Enteric Hyperoxaluria
Brief Title: Safety and Tolerability of SYNB8802 in Healthy Adult Volunteers and Adult Subjects With Enteric Hyperoxaluria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Synlogic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SYNB8802-CP-001
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Healthy; Enteric Hyperoxaluria

STUDY DESIGN:
Intervention Model Description: Part 1 - randomized, placebo-controlled multiple-dose escalation Part 2 - randomized, placebo-controlled crossover
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind (Sponsor-open)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- MAD HV: SYNB8802 (1 x 10^11 live cells) (Experimental): HV subjects receive SYNB8802 (1 x 10^11 live cells) TID for 5 days in the MAD study (Part 1).
  Interventions: Drug: SYNB8802
- MAD HV: SYNB8802 (3 x 10^11 live cells) (Experimental): HV subjects receive SYNB8802 (3 x 10^11 live cells) TID for 5 days in the MAD study (Part 1).
  Interventions: Drug: SYNB8802
- MAD HV: SYNB8802 (1 x 10^12 live cells) (Experimental): HV subjects receive SYNB8802 (1 x 10^12 live cells) TID for 5 days in the MAD study (Part 1).
  Interventions: Drug: SYNB8802
- MAD HV: SYNB8802 (optional cohort 1) (Experimental): HV subjects receive SYNB8802 (at a dose to be determined based on the data from the first 3 cohorts) TID for 5 days in the MAD study (Part 1).
  Interventions: Drug: SYNB8802
- MAD HV: SYNB8802 (optional cohort 2) (Experimental): HV subjects receive SYNB8802 (at a dose to be determined based on the data from the first 3 cohorts) TID for 5 days in the MAD study (Part 1).
  Interventions: Drug: SYNB8802
- MAD HV: Placebo (Placebo Comparator): HV subjects receive placebo TID for 5 days in the MAD study (Part 1).
  Interventions: Drug: Placebo
- Crossover Arm 1: SYNB8802 crossover to Placebo (Other): In Part 2 subjects will be randomized (1:1) to receive SYNB8802 TID for 6 days and then, following a washout period, receive Placebo TID for 6 days.
  Interventions: Drug: SYNB8802; Drug: Placebo
- Crossover Arm 2: Placebo crossover to SYNB8802 (Other): In Part 2 subjects will be randomized (1:1) to receive Placebo TID for 6 days and then, following a washout period, receive SYNB8802 TID for 6 days.
  Interventions: Drug: SYNB8802; Drug: Placebo

INTERVENTIONS:
Drug: SYNB8802 — SYNB8802 is formulated as a nonsterile solution intended for oral administration
  Arms: Crossover Arm 1: SYNB8802 crossover to Placebo; Crossover Arm 2: Placebo crossover to SYNB8802; MAD HV: SYNB8802 (1 x 10^11 live cells); MAD HV: SYNB8802 (1 x 10^12 live cells); MAD HV: SYNB8802 (3 x 10^11 live cells); MAD HV: SYNB8802 (optional cohort 1); MAD HV: SYNB8802 (optional cohort 2)
Drug: Placebo — In order to maintain study blinding, matching placebo in identical packaging will be manufactured using an inactive powder
  Arms: Crossover Arm 1: SYNB8802 crossover to Placebo; Crossover Arm 2: Placebo crossover to SYNB8802; MAD HV: Placebo

SUMMARY:
This Phase 1a/b, first-in-human, multiple dose-escalation, randomized, double-blinded, placebo-controlled study is evaluating SYNB8802 in healthy volunteers (HV) and subjects diagnosed with enteric hyperoxaluria (EH). Eligible subjects receive investigational product (IP) and undergo safety monitoring, evaluations, and subsequent follow-up after IP administration.

In Part 2, all evaluations and assessments throughout this study may be conducted either at the clinical site or by a home healthcare professional at an alternative location (e.g., EH patient's home, hotel).

DETAILED DESCRIPTION:
This study is evaluating the safety, tolerability, kinetics, and pharmacodynamics of SYNB8802 within the following 2 study parts:

Part 1 is an inpatient, placebo-controlled, multiple ascending dose (MAD) study in HV male and female subjects in up to 5 dose cohorts (6 treated: 3 placebo) for 5 days of dosing to identify the maximum tolerated dose (MTD).

Part 2 is a placebo-controlled crossover study in up to 20 adult male and female subjects with EH secondary to Roux-en-Y bariatric surgery. Subjects will be randomized to receive either SYNB8802 (at or below the MTD from Part 1) or placebo for six days before crossing over to receive either placebo or SYNB8802 for another six days, respectively. This part of the study has been designed with the flexibility of being able to be conducted either at the clinical site or by a home healthcare professional at an alternative location (e.g., patient's home, hotel).

ELIGIBILITY:
Part 1 Inclusion Criteria:

1. Age ≥ 18 to ≤ 64 years.
2. Body mass index (BMI) 18.5 to 28 kg/m2.
3. Able and willing to voluntarily complete the informed consent process.
4. Available for and agree to all study procedures, including feces, urine, and blood collection and adherence to diet control, inpatient monitoring, follow-up visits, and compliance with all study procedures.
5. Male subjects who are sexually abstinent or surgically sterilized (vasectomy), or those who are sexually active with a female partner(s) and agree to use an acceptable method of contraception (such as a condom with spermicide) combined with an acceptable method of contraception for their non-pregnant female partner(s) (as defined in Inclusion Criterion # 6) after informed consent, throughout the study, and for a minimum of 3 months after the last dose of IMP, and who do not intend to donate sperm in the period from Screening until 3 months following administration of the investigational medical product.
6. Female subjects who meet 1 of the following:

   1. Woman of childbearing potential (WOCBP) must have a negative pregnancy test (human chorionic gonadotropin) at Screening and at baseline prior to the start of IMP and must agree to use acceptable method(s) of contraception, combined with an acceptable method of contraception for their male partner(s) (as defined in Inclusion Criterion # 5) after informed consent, throughout the study and for a minimum of 3 months after the last dose of IMP. Acceptable methods of contraception include hormonal contraception, hormonal or non-hormonal intrauterine device, bilateral tubal occlusion, complete abstinence, vasectomized partner with documented azoospermia 3 months after procedure, diaphragm with spermicide, cervical cap with spermicide, vaginal sponge with spermicide, or male or female condom with or without spermicide.
   2. Premenopausal woman with at least 1 of the following:

   i. Documented hysterectomy ii. Documented bilateral salpingectomy iii. Documented bilateral oophorectomy iv. Documented tubal ligation/occlusion v. Sexual abstinence is preferred or usual lifestyle of the subject c. Postmenopausal women (12 months or more amenorrhea verified by follicle- stimulating hormone [FSH] assessment and over 45 years of age in the absence of other biological or physiological causes).

Part 1 Exclusion Criteria:

1. Acute or chronic medical (including COVID-19 infection), surgical, psychiatric, or social condition or laboratory abnormality that may increase subject risk associated with study participation, compromise adherence to study procedures and requirements, or may confound interpretation of study safety or PD results and, in the judgment of the investigator, would make the subject inappropriate for enrollment.
2. Body mass index (BMI) < 18.5 or > 28 kg/m2.
3. Oxalobacter formigenes carrier.
4. Pregnant (self or partner), or lactating.
5. Unable or unwilling to discontinue vitamin C supplementation for the study duration.
6. History of or current immunodeficiency disorder including autoimmune disorders and human immunodeficiency virus (HIV) antibody positivity.
7. Hepatitis B surface antigen positivity (subjects with hepatitis B surface antibody positivity and hepatitis B core antibody positivity are not excluded, provided that the hepatitis B surface antigen is negative).
8. Hepatitis C antibody positivity, unless a hepatitis C virus ribonucleic acid test is performed, and the result is negative.
9. History of febrile illness, confirmed bacteremia, or other active infection deemed clinically significant by the investigator within 30 days prior to the anticipated first dose of IMP.
10. History of (within the past month) passage of 3 or more loose stools per day; where 'loose stool' is defined as a Type 6 or Type 7 on the Bristol Stool Chart (see Appendix 1: Bristol Stool Chart).
11. History of kidney stones, renal or pancreatic disease.
12. GI disorder (including inflammatory or irritable bowel disorder of any grade and surgical removal of bowel sections) that could be associated with increased UOx levels.
13. Active or past history of GI bleeding within 60 days prior to the Screening Visit as confirmed by hospitalization-related event(s) or medical history of hematemesis or hematochezia.
14. Intolerance of or allergic reaction to EcN, esomeprazole or PPIs in general, or any of the ingredients in SYNB8802 or placebo formulations.
15. Any condition (e.g., celiac disease, gastrectomy, bypass surgery, ileostomy), prescription medication, or over-the-counter product that may possibly affect absorption of medications or nutrients.
16. Currently taking or plans to take any type of systemic (e.g., oral or intravenous) antibiotic within 30 days prior to Day 1 through the final day of inpatient monitoring. Exception: topical antibiotics are allowed.
17. Major surgery (an operation upon an organ within the cranium, chest, abdomen, or pelvic cavity) or inpatient hospital stay within the past 3 months prior to Screening.
18. Planned surgery, hospitalizations, dental work, or interventional studies between Screening and last anticipated visit that might require antibiotics.
19. Taking or planning to take probiotic supplements (enriched foods excluded) within 30 days prior to Day -1 and for the duration of participation and follow-up.
20. Dependence on alcohol or drugs of abuse.
21. Administration or ingestion of an investigational drug within 30 days or 5 half-lives, whichever is longer, prior to Screening Visit; or current enrollment in an investigational study.
22. Screening laboratory parameters (e.g., chemistry panel, hematology, coagulation) and ECG outside of the normal limits based on standard ranges, or as defined in the table below, or as judged to be clinically significant by the investigator. A single repeat evaluation is acceptable.

Part 2 Inclusion Criteria:

1. Age ≥ 18 to ≤ 74 years.
2. Able and willing to voluntarily complete the informed consent process.
3. Available for and agree to all study procedures, including feces, urine, and blood collection and adherence to diet control, follow-up visits, and compliance with all study procedures.
4. Enteric hyperoxaluria secondary to Roux-en-Y bariatric surgery (at least 12 months post-surgery).
5. Urinary oxalate ≥ 70 mg/24 hours (mean of at least 2 urine collections during Screening).
6. Male subjects who are sexually abstinent or surgically sterilized (vasectomy), or those who are sexually active with a female partner(s) and agree to use an acceptable method of contraception (such as condom with spermicide) combined with an acceptable method of contraception for their non-pregnant female partner(s) (as defined in Inclusion Criterion # 7) after informed consent, throughout the study, and for a minimum of 3 months after the last dose of IMP, and who do not intend to donate sperm in the period from Screening until 3 months following administration of the investigational medical product.
7. Female subjects who meet 1 of the following:

   1. Woman of childbearing potential (WOCBP) must have a negative pregnancy test (human chorionic gonadotropin) at Screening and at baseline prior to the start of IMP and must agree to use acceptable method(s) of contraception, combined with an acceptable method of contraception for their male partner(s) (as defined in Inclusion Criterion # 6) after informed consent, throughout the study and for a minimum of 3 months after the last dose of IMP. Acceptable methods of contraception include hormonal contraception, hormonal or non-hormonal intrauterine device, bilateral tubal occlusion, complete abstinence, vasectomized partner with documented azoospermia 3 months after procedure, diaphragm with spermicide, cervical cap with spermicide, vaginal sponge with spermicide, or male or female condom with or without spermicide.
   2. Premenopausal woman with at least 1 of the following:

   i. Documented hysterectomy ii. Documented bilateral salpingectomy iii. Documented bilateral oophorectomy iv. Documented tubal ligation/occlusion v. Sexual abstinence is preferred or usual lifestyle of the subject c. Postmenopausal women (12 months or more amenorrhea verified by FSH assessment and over 45 years of age in the absence of other biological or physiological causes).
8. Screening laboratory evaluations (e.g., chemistry panel, complete blood count with differential, prothrombin time [PT]/activated partial thromboplastin time [aPTT], urinalysis) and electrocardiogram (ECG) must be within normal limits or judged to be not clinically significant by the investigator.

Part 2 Exclusion Criteria:

1. Acute or chronic medical (including COVID-19 infection), surgical, psychiatric, or social condition or laboratory abnormality that may increase subject risk associated with study participation, compromise adherence to study procedures and requirements, or may confound interpretation of study safety or PD results and, in the judgment of the investigator, would make the subject inappropriate for enrollment.
2. Acute renal failure or eGFR < 45 mL/min/1.73 m2. A single repeat evaluation is acceptable.
3. Unable or unwilling to discontinue vitamin C supplementation for the study duration.
4. Diagnosis of primary hyperoxaluria or any other cause of hyperoxaluria.
5. Oxalobacter formigenes carrier.
6. Pregnant (self or partner), or lactating.
7. Currently taking or plans to take any type of systemic (e.g., oral or intravenous) antibiotic within 30 days prior to Day 1 through the final safety assessment. Exception: topical antibiotics are allowed.
8. Major surgery (an operation upon an organ within the cranium, chest, abdomen, or pelvic cavity) or inpatient hospital stay within the past 3 months prior to Screening.
9. Planned surgery, hospitalizations, dental work, or interventional studies between Screening and last anticipated visit.
10. Taking or planning to take probiotic supplements (enriched foods excluded) within 30 days prior to Day -1 and for the duration of participation.
11. Intolerance of or allergic reaction to EcN, esomeprazole or PPIs in general, or any of the ingredients in SYNB8802 or placebo formulations.
12. Dependence on alcohol or drugs of abuse.
13. History of or current immunodeficiency disorder including autoimmune disorders and HIV antibody positivity.
14. Hepatitis B surface antigen positivity (subjects with hepatitis B surface antibody positivity and hepatitis B core antibody positivity are not excluded, provided that the hepatitis B surface antigen is negative).
15. Hepatitis C antibody positivity, unless a hepatitis C virus ribonucleic acid test is performed, and the result is negative.
16. Administration or ingestion of an investigational drug within 30 days or 5 half-lives, whichever is longer, prior to Screening Visit; or current enrollment in an investigational study.
17. History of bacteremia within 30 days prior to the anticipated first dose of IMP.
18. History of inflammatory bowel disease.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Number of Subjects With Treatment-Emergent Adverse Events | 33 Days
  Toxicity is graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. Adverse events (AEs) are reported based on clinical laboratory tests, vital signs, physical examinations, electrocardiograms, and any other medically indicated assessments from the time informed consent is signed through the end of the safety follow-up period.
  AEs are considered to be treatment emergent (TEAE) if they occur or worsen in severity after the first dose of study treatment. TEAEs are considered treatment-related if relationship to study drug is possibly related, probably related, or definitely related.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Urological Associates of Southern Arizona (open to remote participation), Tucson, Arizona
  - Genesis Clinical Research, Tampa, Florida
  - Knoxville Kidney Center, Knoxville, Tennessee
  - PRA Health Sciences, Salt Lake City, Utah